CLINICAL TRIAL: NCT01404468
Title: Effect of Lidocaine Phonophoresis on Sensory Blockade: Pulsed or Continuous Mode of Therapeutic Ultrasound?
Brief Title: The Phonophoresis of Lidocaine Gel and Its Effect on Sensory Blockage
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: rehabilitation school boss, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 84-7.33
Record Dates: First submitted 2011-07-21; First posted 2011-07-28 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-03

CONDITIONS: Pain; Impairment, Light Touch Sensation
MeSH Terms: conditions — Pain; Somatosensory Disorders | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pulsed (Active Comparator)
  Interventions: Device: pulsed ultrasound device with lidocaine
- control (Sham Comparator)
  Interventions: Other: off device
- continuous (Active Comparator)
  Interventions: Device: continuous ultrasound device with lidocaine

INTERVENTIONS:
Device: pulsed ultrasound device with lidocaine — Lidocaine (approximately 2 cc) was administered transdermally using a transducer (pulsed ultrasound)
  Other Names: lidocainegel(Akron,Inc.,Lake Forest,CA,USA); ultrasound(Enraf,Sonopuls 434,Netherlands)
  Arms: pulsed
Other: off device — off device with Lidocaine (approximately 2 cc) was administered transdermally
  Other Names: ultrasound(Enraf,Sonopuls 434,Netherlands)
  Arms: control
Device: continuous ultrasound device with lidocaine — Lidocaine (approximately 2 cc) was administered transdermally using a transducer (continuous ultrasound )
  Other Names: lidocaine gel(Akron, Inc.,Lake Forest,CA,USA); ultrasound (Enraf,Sonopuls 434,Netherlands)
  Arms: continuous

SUMMARY:
The optimisation of drug absorption through skin is of great value in modern therapy.Phonophoresis is the use of therapeutic ultrasound to increase percutaneous drug absorption. However,few studies have compared pulsed and continuous modes of therapeutic ultrasound.This study compared these two modes by investigating the effect of lidocaine phonophoresis on sensory blockade.

Ninety-three healthy volunteers, assigned at random to one of three ultrasound groups:pulsed(ultrasound+lidocaine),continuous(ultrasound+lidocaine)and control(sham ultrasound+lidocaine).

Lidocaine was administered transdermally using a transducer.Two point discrimination, touch and maximum pain thresholds were assessed before and after the intervention in each group.

Pulsed ultrasound with topical lidocaine gel induced greater anaesthetic effect compared with continuous ultrasound with topical lidocaine gel and lidocaine application alone. The mechanical properties of pulsed ultrasound appear to be responsible for greater drug penetration.

DETAILED DESCRIPTION:
Lidocaine is a common local anaesthetic drug that is used topically to relieve pain,itching and burning, and also for minor surgery.However,its application via this conductive method,has been confined to surface anaesthesia because it seems that it is not possible to have a deep transmission with local drug massage, without injection or systematic administration.On the other hand,the injection of lidocaine can lead to tissue injury and pain,and its use is not advised in children. Phonophoresis is one of the common procedures for reducing these problems. Therefore, the main aim of this study was to compare the two modes of therapeutic ultrasound by assessing the effect of lidocaine gel phonophoresis on percutaneous absorption and sensory blockade.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 25 years

Exclusion Criteria:

* individuals who had a disease that could affect the experiment, such as systemic disease,impairment of the sensory system(e.g.neuropathy,diabetes),cardiovascular disorders(e.g. increased blood pressure),pain due to an injury to the upper extremity,tumours,malignant and precancerous tissue,acute infection and broken skin in the area; and individuals taking medication to relieve disease symptoms were excluded

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Two-point discrimination,touch and maximum pain thresholds | imediately after finishing the application of ultrasound (5 minutes after intervention)

CONTACTS AND LOCATIONS:
Overall Officials: samaneh ebrahimi, PhD student, Principal Investigator — PhD student in shiraz university of medical sciences
Locations (1):
- Samaneh Ebrahimi, Shiraz, Fars, Iran

REFERENCES:
- [Result] Ebrahimi S, Abbasnia K, Motealleh A, Kooroshfard N, Kamali F, Ghaffarinezhad F. Effect of lidocaine phonophoresis on sensory blockade: pulsed or continuous mode of therapeutic ultrasound? Physiotherapy. 2012 Mar;98(1):57-63. doi: 10.1016/j.physio.2011.01.009. PMID 22265386